CLINICAL TRIAL: NCT06472427
Title: The Acute Effect of (R)-1,3-butanediol Ingestion on Post-exercise Skeletal Muscle Angiogenesis in Healthy Adults Under Normoxic and Hypoxic Conditions.
Brief Title: The Effect of Butanediol Ingestion on Skeletal Muscle Angiogenesis in Hypoxia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Chiel Poffé, Principal Investigator, KU Leuven
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: S68402
Record Dates: First submitted 2024-05-30; First posted 2024-06-25 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Ketosis; Hypoxia; Angiogenesis
Keywords: Exercise; Recovery; Living high training low
MeSH Terms: conditions — Ketosis; Hypoxia; Motor Activity | interventions — Ketones

STUDY DESIGN:
Intervention Model Description: 1 session with normoxic post-exercise recovery, supplemented with placebo (NPL)
  1 session with normoxic post-exercise recovery, supplemented with ketones (NKE)
  1 session with hypoxic post-exercise recovery, supplemented with placebo (HPL)
  1 session with hypoxic post-exercise recovery, supplemented with ketones (HKE)
Who Masked: Participant, Investigator
Masking Description: Both participants and investigators actively parttaking in the study are blinded.
  Participants are misinformed that all sessions will be hypoxic, in order to prevent identification of normoxic vs hypoxic conditions. Therefore, participants are also misinformed about the supplements, where they think they will receive 4 different compositions of ketones.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- 1 session with normoxic post-exercise recovery, supplemented with placebo (NPL) (Placebo Comparator): Normoxic training, followed by normoxic recovery with placebo supplements
  Interventions: Dietary Supplement: Normoxic recovery and placebo (NPL)
- 1 session with normoxic post-exercise recovery, supplemented with ketones (NKE) (Experimental): Normoxic training, followed by normoxic recovery with ketone supplements
  Interventions: Dietary Supplement: Normoxic recovery and ketones (NKE)
- 1 session with hypoxic post-exercise recovery, supplemented with placebo (HPL) (Experimental): Normoxic training, followed by hypoxic (simulated altitude of 3000m) recovery with placebo supplements
  Interventions: Dietary Supplement: Hypoxic recovery and placebo (HPL)
- 1 session with hypoxic post-exercise recovery, supplemented with ketones (HKE) (Experimental): Normoxic training, followed by hypoxic (simulated altitude of 3000m) recovery with ketone supplements
  Interventions: Dietary Supplement: Hypoxic recovery and ketones (HKE)

INTERVENTIONS:
Dietary Supplement: Normoxic recovery and placebo (NPL) — Altitude: sea level Dietary supplement: placebo. Water: 98.3% w/w Bitter flavour type: 0.7% w/w Monk fruit extract: 0.04% w/w Tasteva: 0.03% w/w Citric acid: 0.6% w/w Flavor blend: 0.02% w/w Bitter masking flavour: 0.2% w/w Passion fruit flavour: 0.005% w/w
  Arms: 1 session with normoxic post-exercise recovery, supplemented with placebo (NPL)
Dietary Supplement: Normoxic recovery and ketones (NKE) — Altitude: sea level Dietary supplement: Commercially available Ketone-IQ butanediol drink R-1,3-butanediol: 28.6% w/v in water
  Arms: 1 session with normoxic post-exercise recovery, supplemented with ketones (NKE)
Dietary Supplement: Hypoxic recovery and placebo (HPL) — Altitude: 3,000m (simulated) Dietary supplement: placebo. Water: 98.3% w/w Bitter flavour type: 0.7% w/w Monk fruit extract: 0.04% w/w Tasteva: 0.03% w/w Citric acid: 0.6% w/w Flavor blend: 0.02% w/w Bitter masking flavour: 0.2% w/w Passion fruit flavour: 0.005% w/w
  Arms: 1 session with hypoxic post-exercise recovery, supplemented with placebo (HPL)
Dietary Supplement: Hypoxic recovery and ketones (HKE) — Altitude: 3,000m (simulated) Dietary supplement: Commercially available Ketone-IQ butanediol drink R-1,3-butanediol: 28.6% w/v in water
  Arms: 1 session with hypoxic post-exercise recovery, supplemented with ketones (HKE)

SUMMARY:
This study specifically aims to elucidate the effects of intermittent exogenous ketosis (IEK) as well as hypoxia on muscular pro-angiogenic factors- after a 60-min HIIT bout in normoxia. Moreover, blood and muscle oxygenation status, as well as peripheral blood flow and cognitive function will be assessed.

DETAILED DESCRIPTION:
After an exercise bout, angiogenesis is incredibly important in the recovery process as an increased number of capillaries enables higher metabolite transport to and from the working muscle. Often, a training strategy consists of living-high (sleeping at -stimulated- altitude) and training low (training at sea level). A decreased oxygen availability, also known as hypoxia, however poses an additional stress on the human body, potentially compromising the overall training efficiency. Ketones are recently found to increase angiogenesis in response to overload training (increased skeletal muscle capillarization and VEGF content) and to increase serum EPO concentrations. Therefore, the investigators want to evaluate the isolated and interactive effects of both ketones and hypoxia on post-exercise recovery and factors implicated in skeletal muscle angiogenesis, after training in normoxia. Moreover, a performance test will be performed after 7h of hypoxic or normoxic recovery by means of a simulated 15 min all-out time trial. During the 7h post-exercise window, biological samples are collected (muscle biopsies, venous blood samples, urine, capillary blood samples). Moreover, blood and muscle oxygenation, peripheral blood flow and cognitive function are assessed at regular timepoints.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be obtained prior to any experimental procedures
2. Biological male or biological females using oral contraception between 18 and 35 years old
3. Recreational or competitive cyclists performing regularly cycling training sessions with an average training volume of more than 6 hours per week
4. Good health status confirmed by a medical screening
5. Body Mass Index (BMI) between 18 and 25 kg/m2

Exclusion Criteria:

1. Any kind of injury/pathology that is a contra-indication for hypoxic exposure and/or to perform high-intensity exercise, evaluated by a sport medical screening
2. Intake of any medication or nutritional supplement that is known to affect exercise or performance. Intake will be assessed during recruitment and the sport medical screening.
3. Intake of analgesics, anti-inflammatory agents, or supplementary anti-oxidants, within two weeks of study participation.
4. Recent residence or training under hypoxia; more than 7 days exposure to altitude > 1500 m during the 3 months preceding the study.
5. Blood donation within 3 months of study participation.
6. Habitual smoking
7. Pre-existing, diagnosed psychiatric conditions or anxiety
8. Females that are pregnant or are planning to be pregnant before the end of the study (end of May 2024)
9. Depression or anxiety as assessed by the Beck Depression Inventory 25 (Appendix 2) and Beck Anxiety Inventory 26 (Appendix 3). Only a score in the range of 'normal ups and downs' (score 1-10) for depression or 'minimal anxiety' (score 0-7) for anxiety are tolerated.
10. History of addiction or excessive caffeine/alcohol consumption assessed by a questionnaire (Appendix 4).
11. Any other reason that might pose undue risk to the participant, or introduce bias into the study outcomes, at the discretion of the research team.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Post-exercise muscle VEGF mRNA expression | Muscle biopsies are collected 10 minutes after the end of training as well as 3 hours later.
  Measured using PCR on collected muscle biopsies
Post-exercise serum EPO concentrations | Venous blood samples are collected 10 minutes after the end of training as well as 3 hours, 5 hours and 7 hours later.
  Measured using ELISA on collected serum samples

SECONDARY OUTCOMES:
Change in muscular VEGF concentration | Muscle biopsies are collected 10 minutes after the end of training as well as 3 hours later.
  Measured using Western Blotting on muscle biopsies
Change in serum VEGF concentration | Venous blood samples are collected immediately (5 minutes) after the end of training, as well as 3hours, 5hours and 7hours later..
  Measured using ELISA on collected serum samples
Change in blood oxygenation | Continuously measured starting 30 minutes after the end of exerciseuntil 7.5 hours later
  Measured using pulse oximetry with a sensor on the forehead
Change in skeletal muscle oxygenation | Measured during resting measurements performed 30 minutes, 3hours and 30minutes as well as 6hours and 30minutes after the end of training.
  Measured using NIRS with a sensor on the belly of the m. vastus lateralis (skeletal muscle)
Change in peripheral blood flow | Measured during resting measurements performed 30 minutes, 3hours and 30minutes as well as 6hours and 30minutes after the end of the training
  Measured using duplex ultrasonography
Exercise performance | Performed 7hours and 30minutes after the end of training
  Measured as the average power output (W) during a 15 minutes all-out time trial

OTHER OUTCOMES:
Change in citrate synthase as a marker of mitochondrial density | Muscle biopsies are collected 10 minutes after the end of training as well as 3 hours later.
  Measured using an enzymatic essay

CONTACTS AND LOCATIONS:
Overall Officials: Chiel Poffé, Principal Investigator — KU Leuven
Locations (1):
- KU Leuven, Leuven, Vlaams-Brabant, Belgium